CLINICAL TRIAL: NCT00363727
Title: A Two Year Phase IIIb Randomised, Multicenter, Double-blind, SINEMET Controlled, Parallel Group, Flexible Dose Study, to Assess the Effectiveness of Controlled Release Ropinirole add-on Therapy to L-dopa at Increasing the Time to Onset of Dyskinesia in Parkinson's Disease Subjects.
Brief Title: Onset Motor Complications Using REQUIP CR (Ropinirole Controlled-release) As Add-on Therapy To L-dopa In Parkinson's
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 101468/228
Record Dates: First submitted 2006-08-07; First posted 2006-08-15 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Parkinson's Disease; Parkinson Disease; Dyskinesias
Keywords: dyskinesia; SINEMET; Parkinson's disease; controlled release ropinirole
MeSH Terms: conditions — Parkinson Disease; Dyskinesias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ropinirole controlled-release (REQUIP CR) for RLS

SUMMARY:
This study evaluates how effective a new formulation of a marketed drug is in increasing the time to onset of dyskinesia (abnormal twisting, writhing movements) in patients with Parkinson's Disease who have been taking levodopa for less than 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Must be on 600mg or less of levodopa therapy for two years or less.
* Must be on a stable dose of levodopa therapy for at least 4 weeks prior to screening.

Exclusion Criteria:

* Current or past history of Dyskinesia.
* State of dementia or have a MMSE score < 26 at screening.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2003-12; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with time to onset of dyskinesia of treatment over 104 weeks (2 years) | Up to 2 Years
  Median time to dyskinesia could not be estimated by Kaplan-Meier methods because of the small number of events; however, number of participants with dyskinesia requiring days from the date of randomization (Day 1) to the date at which a participant has the event of interest were reported

SECONDARY OUTCOMES:
Change from Baseline (Day 1) in united PD rating scale (UPDRS) activities of daily living (ADL) score (Part II) at Week 28 and 104 | At Weeks 28 and 104
  UPDRS assessments were conducted within a window of at least 2 hours after the previous L-dopa dose and prior to the next scheduled L-dopa dose. Participants might had been evaluated in either the "on" or "off" states and the summaries of the UPDRS motor score at each visit were produced separately for each state. Change from Baseline is the score at indicated time point minus the score at Baseline. This scale is a clinician-based rating scale used to measure motor impairments and disability. The UPDRS assesses 6 features of Parkinson's disease (PD) impairment that are evaluated using a combination of data collected by interview and participant examination. Part II had 13 questions with ADL scale ranging from 0-52 with 0 indicating no complications and higher scores indicating more severe complications. Week 104 are the records with last observation carries forward (LOCF).
Change from Baseline (Day 1) UPDRS motor score (UPDRS Part III) over period at Week 28 and Week 104 | Baseline (Day 1), Week 28, and Week 104
  UPDRS assessments were conducted within a window of at least 2 hours after the previous L-dopa dose and prior to the next scheduled L-dopa dose. Participants might had been evaluated in either the "on" or "off" states and the summaries of the UPDRS motor score at each visit were produced separately for each state. Change from Baseline is the score at indicated time point minus the score at Baseline. This scale is a clinician-based rating scale used to measure motor impairments and disability. The UPDRS assesses 6 features of Parkinson's disease (PD) impairment that are evaluated using a combination of data collected by interview and participant examination. Part III had 14 questions with ADL scale ranging from 0-56 with 0 indicating no complications and higher scores indicating more severe complications.
Number of participants with symptoms of dyskinesia over period | Upto week 106
  Responses to dyskinesia-related items on the Baseline UPDRS Part IV (Day 1) were analyzed. Part IV of the UPDRS includes 11 questions, four scored with 5-point Likert scales on which higher scores represent more severe complications.
Change from Baseline (Day 1) in fatigue score using epworth sleepiness scale (ESS) over period | Baseline (Day 1) and up to Week 104
  ESS is a brief self-administered questionnaire which asks the participant to rate on a scale of 0-3 ("would never doze" to "high chance of dozing") and was rated relative to the previous week. The scale thus indicated participants to retrospectively characterize their usual behavior in a variety of situations which were more or less soporific. The ESS score is the sum of the 8 item scores and can range from 0-24. This scale was to be administered at Baseline (Day 1), Week 28, Week 52, Week 76, Week 104. Week 104 analysis was based on LOCF. Change from Baseline (Day 1) is the value at indicated time point minus the Baseline value.
Percentage of participants with reduced PD symptom control up to 96 weeks | Up to Week 96
  Time to onset of motor fluctuations (for purposes of this study this is defined as Onset of Wearing Off) over period was analyzed as a measure of number of participants with Reduced Parkinson's Disease Symptom Control. 'Yes' response to the question "Did the participant experience a reduction in Parkinson's disease symptom control within four hours of the dose of L-dopa or the study drug " was analyzed and number of participants showing the response were recorded. The dose was adjusted as per the symptom control. No more data was reported post 96 weeks.
Percentage of participants with a score of "much improved" or "very much improved" on the clinical global impression of improvement (CGI -I) up to 52 weeks | Up to 52 weeks
  The CGI-I scale allows the Investigator to rate the participant's total improvement since beginning the treatment (Baseline/ Day 1). The scale was rated from 1-7 (1="very much improved", 7= "very much worse") from Week 1 onwards will the first year (and at early withdrawal, if applicable).
Mean change from Baseline (Day 1) in PD quality of life score (PDQ39) scale over period | Up to 104 weeks
  Week 104 analysis was LOCF analysis. Change from Baseline (Day 1) is the value at indicated time point minus the value at Baseline.
Mini mental status examination (MMSE) score status at screening and Week 104 | Screening and Week 104
  MMSE is a brief, easily administered mental status examination which is highly reliable and a valid instrument for detecting and tracking the progression of cognitive impairment associated with neurogenerative diseases. The MMSE scale consists of 11 items, with total maximum items scores ranging from 1 to 5. The total maximum score for the MMSE is calculated as the sum of scores for each of the 11 items that is 30, representing the highest level of mental functioning.
Change from Baseline (Day 1) in total score on the beck depression inventory (BDI) over period | Baseline (Day 1) and up to Week 104
  BDI version II (BDI-II) is a 21-item questionnaire that is completed by the participant (the recommended method of use is by assisted self-rating). The BDI included 21 ordered groups of statements from which participants selected the most appropriate description for themselves. Nineteen groups allow a choice from four statements and two sets allow a choice from seven statements. Each group of statements was scored based on the relative severity of the statement chosen, with higher scores representing greater severity. The total BDI score is the sum of scores from the 21 statement groups; total ranging from 0-69, with high values representing the more severe depression.
Change from Baseline (Day 1) in night-time quality of sleep scores of the PD sleep scale (PDSS) over period | Week 28, 52, 76, and 104
  PDSS scale consists of a series of 15 visual analogue scales (VAS) addressing commonly reported symptoms associated with sleep disturbance in PD. The participant or caregiver (by proxy) completed the scale based on their experiences in the past week. The severity of symptoms is reported by marking a cross on each 10 centimeters (cm) VAS line (labeled from worst to best state). Responses were quantified by measuring the distance along each line where the cross was placed. Thus, scores for each item ranged from 0 (symptom severe and always experienced) to 10 (symptom free). The maximum cumulative score for the PDSS was 150 (participant is free of all symptoms); total score was made of cumulative distance scores from fifteen 10 cm lines. Change from Baseline (Day 1) is the value at indicated time point minus the baseline value. Analysis at Week 104 was LOCF observation.
Percentage of participants of genes variants of interest with and without dyskinesia over period | Up to Week 104
  The percentage of randomized participants who consented to genotype sampling and for whom a blood sample was actually collected were summarized; however, no conclusions were drawn, since the pharmacogenetic analysis of the dyskinesia events was not undertaken.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (64):
- United States (64):
  - GSK Investigational Site, Anniston, Alabama
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Sun City, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Oxnard, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Boulder, Colorado
  - GSK Investigational Site, Danbury, Connecticut
  - GSK Investigational Site, Newark, Delaware
  - GSK Investigational Site, Boca Raton, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Palm Beach Gardens, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Port Charlotte, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Austell, Georgia
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Hoffman Estates, Illinois
  - GSK Investigational Site, Northbrook, Illinois
  - GSK Investigational Site, Des Moines, Iowa
  - GSK Investigational Site, Kansas City, Kansas
  - GSK Investigational Site, Elkridge, Maryland
  - GSK Investigational Site, South Weymouth, Massachusetts
  - GSK Investigational Site, West Yarmouth, Massachusetts
  - GSK Investigational Site, Bingham Farms, Michigan
  - GSK Investigational Site, Grand Rapids, Michigan
  - GSK Investigational Site, Traverse City, Michigan
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Edison, New Jersey
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Amherst, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Lubbock, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Alexandria, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Roanoke, Virginia
  - GSK Investigational Site, Kirkland, Washington
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Charleston, West Virginia
  - GSK Investigational Site, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] R Watts, K Sethi, R Pahwa, B Adams, N Earl. Ropinirole 24-hour prolonged release delays the onset of dyskinesia Compared with carbidopa/levodopa in patients with Parkinson's disease treated with levodopa. Eur J Neurol. 2007;14 (Issue s1):1-355 .
- [Background] R Watts, K Sethi, R Pahwa, B Adams, N Earl. Ropinirole 24-hour prolonged release delays the onset of dyskinesia compared with carbidopa/levodopa in patients with Parkinson's disease treated with levodopa. Movement Disorders. 2007;22 (Suppl.16):S94/307.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 101468/228 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 101468/228 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 101468/228 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 101468/228 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 101468/228 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 101468/228 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 101468/228 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register